CLINICAL TRIAL: NCT02783950
Title: Genomics in Michigan Impacting Observation or Radiation (G-MINOR)
Brief Title: Genomics in Michigan Impacting Observation or Radiation
Acronym: G-MINOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Michigan Urological Surgery Improvement Collaborative (MUSIC) (Other); GenomeDx Biosciences Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UMCC 2016.020; CU 008 (Other: GenomeDx Biosciences Corp); HUM00110858 (Other: University of Michigan)
Record Dates: First submitted 2016-05-24; First posted 2016-05-26 (Estimated); Results first posted 2021-02-25 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer
Keywords: Genomics; Adjuvant Treatment
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GC (Decipher) Arm (Other): If enrolled during the Genomic Classifier (GC) period, both subjects and their treating physician will be provided GC (Decipher Prostate Cancer Classifier from GenomeDx) and CAPRA-S scores following prostatectomy.
  Interventions: Other: Decipher Prostate Cancer Classifier
- Usual-Care-Based (UC) Arm (No Intervention): If enrolled during the UC period, only the CAPRA-S results will be provided.

INTERVENTIONS:
Other: Decipher Prostate Cancer Classifier — The Decipher test (GenomeDx Biosciences, San Diego, CA) is a genomic test that predicts high grade disease, the probability of metastasis and prostate cancer-specific mortality for men with prostate cancer.
  Other Names: Decipher Post-Op
  Arms: GC (Decipher) Arm

SUMMARY:
To determine the impact of Decipher test results on adjuvant treatment decisions of high-risk post-RP patients with undetectable post-op prostate specific antigen (PSA) compared to clinical factors alone.

DETAILED DESCRIPTION:
This prospective, randomized trial will compare the receipt of adjuvant therapy for high-risk radical prostatectomy (RP) patients who undergo Decipher testing to those who do not. 350 subjects from within the statewide Michigan Urological Surgery Improvement Collaborative (MUSIC) will be randomized to either a Genomic Classifier (Decipher) or Usual-Care-Based (UC) strategy for a period of three months. If enrolled during the Genomic Classifier period, both subjects and their treating physician will be provided Decipher results and CAPRA-S scores. In the UC periods, CAPRA-S scores but not Decipher results will be provided.

The enrollment goal, initially and throughout the study, was to enroll 350 evaluable patients. During the study, the target accrual goal was raised to 550 patients to allow more flexibility among sites to achieve the enrollment goal of 350 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients who have undergone radical prostatectomy
* PSA < 0.1 ng/ml at enrollment
* At least one of the following:

  * pT3 (seminal vesicle invasion or extraprostatic extension), or
  * Positive surgical margins
* Radical prostatectomy within one year of enrollment

Exclusion Criteria:

* Individuals who have any of the following will not be eligible to participate:

  * Have regional or distant metastatic disease
  * Received any radiation or hormone therapy (neo-adjuvant, adjuvant, or salvage)
  * Node positive

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2024-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Morgan, MD, Principal Investigator — University of Michigan; Michael Cher, MD, Principal Investigator — Wayne State University
Locations (13):
- United States (13):
  - University of Michigan Hospital and Health Systems, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Urologic Consultants, Grand Rapids, Michigan
  - Urology Associates of Grand Rapids, Grand Rapids, Michigan
  - Michigan Urological Clinic, Grand Rapids, Michigan
  - Spectrum Health Medical Group- Urology, Grand Rapids, Michigan
  - Urology Surgeons, PC, Grand Rapids, Michigan
  - Comprehensive Medical Center, PLLC, Royal Oak, Michigan
  - Tri-City Urology, Saginaw, Michigan
  - Bay Area Urology Associates, PC, Traverse City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - IHA Urology at St. Joe's Ann Arbor, Ypsilanti, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams G, Gulliford MC, Ukoumunne OC, Eldridge S, Chinn S, Campbell MJ. Patterns of intra-cluster correlation from primary care research to inform study design and analysis. J Clin Epidemiol. 2004 Aug;57(8):785-94. doi: 10.1016/j.jclinepi.2003.12.013. PMID 15485730
- [Background] Badani K, Thompson DJ, Buerki C, Davicioni E, Garrison J, Ghadessi M, Mitra AP, Wood PJ, Hornberger J. Impact of a genomic classifier of metastatic risk on postoperative treatment recommendations for prostate cancer patients: a report from the DECIDE study group. Oncotarget. 2013 Apr;4(4):600-9. doi: 10.18632/oncotarget.918. PMID 23592338
- [Background] Buja, A., Hastie, T. J. and Tibshirani, R. J. (1989). Linear smoothers and additive models (with discussion). Annals of Statistics, 17, 453-555.
- [Background] Badani KK, Thompson DJ, Brown G, Holmes D, Kella N, Albala D, Singh A, Buerki C, Davicioni E, Hornberger J. Effect of a genomic classifier test on clinical practice decisions for patients with high-risk prostate cancer after surgery. BJU Int. 2015 Mar;115(3):419-29. doi: 10.1111/bju.12789. Epub 2014 Aug 11. PMID 24784420
- [Background] Campbell, Michael J., and Stephen J. Walters. How to Design, Analyse and Report Cluster Randomised Trials in Medicine and Health Related Research. John Wiley & Sons, 2014.
- [Background] Erho N, Crisan A, Vergara IA, Mitra AP, Ghadessi M, Buerki C, Bergstralh EJ, Kollmeyer T, Fink S, Haddad Z, Zimmermann B, Sierocinski T, Ballman KV, Triche TJ, Black PC, Karnes RJ, Klee G, Davicioni E, Jenkins RB. Discovery and validation of a prostate cancer genomic classifier that predicts early metastasis following radical prostatectomy. PLoS One. 2013 Jun 24;8(6):e66855. doi: 10.1371/journal.pone.0066855. Print 2013. PMID 23826159
- [Background] Heo M, Leon AC. Comparison of statistical methods for analysis of clustered binary observations. Stat Med. 2005 Mar 30;24(6):911-23. doi: 10.1002/sim.1958. PMID 15558576
- [Background] Karnes RJ, Bergstralh EJ, Davicioni E, Ghadessi M, Buerki C, Mitra AP, Crisan A, Erho N, Vergara IA, Lam LL, Carlson R, Thompson DJ, Haddad Z, Zimmermann B, Sierocinski T, Triche TJ, Kollmeyer T, Ballman KV, Black PC, Klee GG, Jenkins RB. Validation of a genomic classifier that predicts metastasis following radical prostatectomy in an at risk patient population. J Urol. 2013 Dec;190(6):2047-53. doi: 10.1016/j.juro.2013.06.017. Epub 2013 Jun 11. PMID 23770138
- [Background] Den RB, Feng FY, Showalter TN, Mishra MV, Trabulsi EJ, Lallas CD, Gomella LG, Kelly WK, Birbe RC, McCue PA, Ghadessi M, Yousefi K, Davicioni E, Knudsen KE, Dicker AP. Genomic prostate cancer classifier predicts biochemical failure and metastases in patients after postoperative radiation therapy. Int J Radiat Oncol Biol Phys. 2014 Aug 1;89(5):1038-1046. doi: 10.1016/j.ijrobp.2014.04.052. Epub 2014 Jul 8. PMID 25035207
- [Background] Cooperberg MR, Davicioni E, Crisan A, Jenkins RB, Ghadessi M, Karnes RJ. Combined value of validated clinical and genomic risk stratification tools for predicting prostate cancer mortality in a high-risk prostatectomy cohort. Eur Urol. 2015 Feb;67(2):326-33. doi: 10.1016/j.eururo.2014.05.039. Epub 2014 Jul 2. PMID 24998118
- [Background] Klein EA, Yousefi K, Haddad Z, Choeurng V, Buerki C, Stephenson AJ, Li J, Kattan MW, Magi-Galluzzi C, Davicioni E. A genomic classifier improves prediction of metastatic disease within 5 years after surgery in node-negative high-risk prostate cancer patients managed by radical prostatectomy without adjuvant therapy. Eur Urol. 2015 Apr;67(4):778-86. doi: 10.1016/j.eururo.2014.10.036. Epub 2014 Nov 12. PMID 25466945
- [Background] Den RB, Yousefi K, Trabulsi EJ, Abdollah F, Choeurng V, Feng FY, Dicker AP, Lallas CD, Gomella LG, Davicioni E, Karnes RJ. Genomic classifier identifies men with adverse pathology after radical prostatectomy who benefit from adjuvant radiation therapy. J Clin Oncol. 2015 Mar 10;33(8):944-51. doi: 10.1200/JCO.2014.59.0026. Epub 2015 Feb 9. PMID 25667284
- [Background] Ross AE, Johnson MH, Yousefi K, Davicioni E, Netto GJ, Marchionni L, Fedor HL, Glavaris S, Choeurng V, Buerki C, Erho N, Lam LL, Humphreys EB, Faraj S, Bezerra SM, Han M, Partin AW, Trock BJ, Schaeffer EM. Tissue-based Genomics Augments Post-prostatectomy Risk Stratification in a Natural History Cohort of Intermediate- and High-Risk Men. Eur Urol. 2016 Jan;69(1):157-65. doi: 10.1016/j.eururo.2015.05.042. Epub 2015 Jun 6. PMID 26058959
- [Background] Yamoah K, Johnson MH, Choeurng V, Faisal FA, Yousefi K, Haddad Z, Ross AE, Alshalafa M, Den R, Lal P, Feldman M, Dicker AP, Klein EA, Davicioni E, Rebbeck TR, Schaeffer EM. Novel Biomarker Signature That May Predict Aggressive Disease in African American Men With Prostate Cancer. J Clin Oncol. 2015 Sep 1;33(25):2789-96. doi: 10.1200/JCO.2014.59.8912. Epub 2015 Jul 20. PMID 26195723
- [Background] Lake S, Kammann E, Klar N, Betensky R. Sample size re-estimation in cluster randomization trials. Stat Med. 2002 May 30;21(10):1337-50. doi: 10.1002/sim.1121. PMID 12185888
- [Background] Michalopoulos SN, Kella N, Payne R, Yohannes P, Singh A, Hettinger C, Yousefi K, Hornberger J; PRO-ACT Study Group. Influence of a genomic classifier on post-operative treatment decisions in high-risk prostate cancer patients: results from the PRO-ACT study. Curr Med Res Opin. 2014 Aug;30(8):1547-56. doi: 10.1185/03007995.2014.919908. Epub 2014 May 15. PMID 24803160
- [Background] Nguyen PL, Shin H, Yousefi K, Thompson DJ, Hornberger J, Hyatt AS, Badani KK, Morgan TM, Feng FY. Impact of a Genomic Classifier of Metastatic Risk on Postprostatectomy Treatment Recommendations by Radiation Oncologists and Urologists. Urology. 2015 Jul;86(1):35-40. doi: 10.1016/j.urology.2015.04.004. PMID 26142578
- [Background] Lobo JM, Dicker AP, Buerki C, Daviconi E, Karnes RJ, Jenkins RB, Patel N, Den RB, Showalter TN. Evaluating the clinical impact of a genomic classifier in prostate cancer using individualized decision analysis. PLoS One. 2015 Apr 2;10(3):e0116866. doi: 10.1371/journal.pone.0116866. eCollection 2015. PMID 25837660
- [Background] Thompson IM, Tangen CM, Paradelo J, Lucia MS, Miller G, Troyer D, Messing E, Forman J, Chin J, Swanson G, Canby-Hagino E, Crawford ED. Adjuvant radiotherapy for pathological T3N0M0 prostate cancer significantly reduces risk of metastases and improves survival: long-term followup of a randomized clinical trial. J Urol. 2009 Mar;181(3):956-62. doi: 10.1016/j.juro.2008.11.032. Epub 2009 Jan 23. PMID 19167731
- [Background] Vickers AJ, Elkin EB. Decision curve analysis: a novel method for evaluating prediction models. Med Decis Making. 2006 Nov-Dec;26(6):565-74. doi: 10.1177/0272989X06295361. PMID 17099194
- [Background] Wu S, Crespi CM, Wong WK. Comparison of methods for estimating the intraclass correlation coefficient for binary responses in cancer prevention cluster randomized trials. Contemp Clin Trials. 2012 Sep;33(5):869-80. doi: 10.1016/j.cct.2012.05.004. Epub 2012 May 22. PMID 22627076
- [Derived] Lewicki P, Jiang R, Singhal U, Daignault-Newton S, Ginsburg K, Borza T, Schipper M, Cher M, Morgan T, Stensland K; Michigan Urological Surgery Improvement Collaborative. How Sticky Are Clinical Trial Interventions? Site-Level Clinical Trial Participation and Differential Post-Trial Use of a Genomic Test. JCO Oncol Pract. 2025 Sep 11:OP2500475. doi: 10.1200/OP-25-00475. Online ahead of print. PMID 40934443
- See also: Website for MUSIC — http://musicurology.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GC (Decipher) Arm | Usual-Care-Based (UC) Arm
Started | 182 | 174
Completed (Includes all patients who were followed for at least 18 months or had an event prior to 18 months) | 175 | 165
Not Completed | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GC (Decipher) Arm | Usual-Care-Based (UC) Arm | Total
Number analyzed (Participants) | 182 | 174 | 356
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (6.5) | 64.6 (6.3) | 64.7 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 182 | 174 | 356
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 149 | 147 | 296
  Unknown or Not Reported | 31 | 25 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 4 | 0 | 4
  Black or African American | 15 | 11 | 26
  White | 140 | 140 | 280
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 22 | 20 | 42
Prostate Specific Antigen [Median (Full Range); unit: ng/ML] | 6.6 [1.1 to 40.2] | 6.0 [1.5 to 30.5] | 6.4 [1.1 to 40.2]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Receive Adjuvant Therapy (Radiation and/or Hormone Therapy)
Description: Adjuvant will be defined as preceding biochemical recurrence (BCR) (i.e.: PSA ≥ 0.2 ng/ml) and within 18 months of radical prostatectomy.
Time Frame: within 18 months of radical prostatectomy
Population: Includes all patients who were followed for at least 18 months or had an event prior to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | GC (Decipher) Arm | Usual-Care-Based (UC) Arm
Number analyzed (Participants) | 175 | 165
Participants | 19 | 12
Statistical Analysis 1: Comparison: GC (Decipher) Arm vs Usual-Care-Based (UC) Arm; Test type: Superiority; p = 0.27, Chi-squared

2. Secondary Outcome: Time (From Randomization) to Adjuvant Treatment Administration
Description: Adjuvant treatment (radiation and/or hormone) is defined as preceding BCR. BCR occurs when prostate specific antigen (PSA) ≥ 0.2 ng/ml.
Time Frame: Up to 18 months post randomization
Population: Population includes patients who had adjuvant treatment
Measure: Median (Full Range); unit: days
Arm/Group | GC (Decipher) Arm | Usual-Care-Based (UC) Arm
Number analyzed (Participants) | 19 | 12
days | 259 [169 to 474] | 233.5 [65 to 501]
Statistical Analysis 1: Comparison: GC (Decipher) Arm vs Usual-Care-Based (UC) Arm; Test type: Superiority; p = 0.70, Wilcoxon Rank Test p-value

3. Secondary Outcome: Time (From Randomization) to Salvage Treatment Administration
Description: Salvage treatment (radiation and/or hormone therapy) is defined as either after BCR or >18 months after surgery in the absence of documented BCR
Time Frame: Up to 5 years post randomization
Reporting Status: Not Posted

4. Secondary Outcome: Time (From Randomization) to Biochemical Recurrence (BCR)
Description: BCR is defined as PSA ≥ 0.2 ng/ml.
Time Frame: Up to 5 years post randomization
Reporting Status: Not Posted

5. Secondary Outcome: Time (From Randomization) to Metastatic Disease (Regional or Distant)
Description: Metastasis is determined based on CT, MRI, bone scan, and/or positron emission tomography (PET) scan
Time Frame: Up to 5 years post randomization
Reporting Status: Not Posted

6. Secondary Outcome: Michigan Urological Surgery Improvement Collaborative (MUSIC) Patient Reported Outcomes (PRO)
Description: Composite Expanded Prostate Cancer Index Composite (EPIC)-26 domain scores for a) urinary irritative function, b) urinary incontinence, and c) sexual function will be measured at baseline and 24 months post-radical prostatectomy. Each of the 3 domains is scaled from 0-100 (higher is better).
Time Frame: Up to 24 months post radical prostatectomy
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | GC (Decipher) Arm | Usual-Care-Based (UC) Arm
All-Cause Mortality (participants affected / at risk) | 2/182 | 0/174
Serious Adverse Events (participants affected / at risk) | 0/182 | 0/174
Other Adverse Events (participants affected / at risk) | 0/182 | 0/174

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/50/NCT02783950/Prot_SAP_000.pdf